CLINICAL TRIAL: NCT01343108
Title: The Impact of Nurses' Emotional Labor on Job Satisfaction and Burnout
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Cheng-I Chu, Tzu Chi University
Other Study IDs: 100001
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Satisfaction
Keywords: Emotional Labor; Burnout; Job Satisfaction; Emotional Intelligence; Job stress; Job involvement
MeSH Terms: conditions — Personal Satisfaction; Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Emotional labor is one of the bases that organizations earn profits. Nursing care needs high emotional labor to offer health care to patients. Among health carers that emphasize a lot on emotional labor, nurses are especially required to include emotional labor as very important parts of their jobs.

DETAILED DESCRIPTION:
This study intends to investigate the association among emotional labor, job satisfaction, and burnout. Furthermore, the moderating effect of job stress , job involvement and emotional intelligence will be studied. The study population includes all nurses (N=18,446) of Taiwan's medical centers. Of which, 20% of randomly selected six medical centers will be delivered a questionnaire in order to further analyze the association of study variables.

The level of emotional labor, burnout, job satisfaction, job stress, job involvement and emotional intelligence of the study samples collected from questionnaires will be analyzed by using descriptive statistics, variance analyses, and SEM techniques in order to understand more the associations among study variables. Results of this study are expected to work as references to improve job satisfaction and decrease the level of burnout of nurses.

ELIGIBILITY:
Inclusion Criteria:

* licensed nurses in the hospitals

Exclusion Criteria:

* part-time nurses
* nurses who work under a year in the hospitals

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: nurses
Sampling Method: Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2011-03; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-I Chu, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, Hualien, Taiwan